CLINICAL TRIAL: NCT02392754
Title: Program for Identification of "Actionable" Atrial Fibrillation (PIAAF): Home-Based Screening for Early Detection of Atrial Fibrillation in Primary Care Patients Aged 75 Years and Older: the SCREEN-AF Randomized Trial
Brief Title: Home-Based Screening for Early Detection of Atrial Fibrillation in Primary Care Patients Aged 75 Years and Older
Acronym: SCREEN-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Stroke Prevention Intervention Network (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Canadian Stroke Network (Other); iRhythm Technologies, Inc. (Industry); Microlife (Industry); University of Leipzig (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SCREEN-AF
Record Dates: First submitted 2015-01-19; First posted 2015-03-19 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation; Hypertension
Keywords: Screening; Atrial Fibrillation; ECG; Primary care
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening (Experimental): The intervention group receives AF screening with a 2-week ambulatory ECG patch monitor (ZIO XT Patch) worn at baseline and again at 3 months, in addition to standard care for 6 months. The intervention group also receives a home BP monitor with automatic AF detection capability to be used twice daily for 2 weeks during the ECG monitoring periods.
  Interventions: Device: Screening: Intervention - Atrial fibrillation screening (ZIO XT ECG monitor, Watch-BP)
- Control (No Intervention): The control group receives standard care for 6 months (including a pulse check and heart auscultation by a physician at 6 months).

INTERVENTIONS:
Device: Screening: Intervention - Atrial fibrillation screening (ZIO XT ECG monitor, Watch-BP) — The intervention group receives AF screening with a 2-week ambulatory ECG patch monitor (ZIO XT Patch) worn at baseline and again at 3 months, in addition to standard care for 6 months. The intervention group also receives a home BP monitor with automatic AF detection capability to be used twice daily for 2 weeks during the ECG monitoring periods.
  Other Names: ZIO XT Patch ambulatory ECG patch monitor; Watch BP-Home A blood pressure monitor
  Arms: Screening

SUMMARY:
Atrial fibrillation (AF) is a major treatable risk factor for stroke, but it may be hard to detect because it is frequently silent and intermittent. New ambulatory cardiac monitoring technologies have the potential to improve early detection of AF. This trial investigates AF screening in primary care patients using the ZIO XT Patch, a wearable adhesive patch monitor that provides continuous ECG recording for up to 14 days, in addition to the WatchBP home blood pressure monitor that has built-in AF screening capability.

DETAILED DESCRIPTION:
SCREEN-AF is an investigator-initiated, multicenter, open-label, two-group randomized controlled trial investigating non-invasive, home-based AF screening. The trial targets patients aged 75 years or older with a history of hypertension and without known AF who would be potential anticoagulant candidates if AF were detected. Eligible participants will be recruited from primary care practices and randomly allocated (1:1) to one of two groups:

* The control group will receive standard care for 6 months (including a pulse check and heart auscultation by a physician at baseline and 6 months).
* The intervention group will undergo ambulatory screening for AF with a 2-week continuous ECG patch monitor worn at baseline and again at 3 months, in addition to standard care for 6 months (including a pulse check and heart auscultation by a physician at baseline and 6 months). The intervention group will also receive a home BP monitor with automatic AF detection capability to be used twice daily for 2 weeks during the ECG monitoring blocks.

The hypothesis is that continuous ambulatory cardiac rhythm monitoring using an adhesive ECG patch monitor will be superior to standard care for AF detection. The overall aim of this research is to establish a practical and cost-effective screening strategy that could be applied in primary care for early detection of AF in patients who would benefit from anticoagulant therapy if AF were detected. The ultimate goal of this primary prevention initiative is to prevent more strokes, and stroke-related deaths, disability, dementia, hospitalizations and institutionalization, through the early detection and treatment of AF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥75 years without known atrial fibrillation or atrial flutter.
2. The participant is clinically in sinus rhythm (both heart auscultation and 30- second pulse palpation have been performed by the enrolling physician and neither detects an irregular rhythm suggestive of atrial fibrillation).
3. History of hypertension requiring antihypertensive medication.
4. Written informed consent from the participant.

Exclusion Criteria:

1. Any previously documented atrial fibrillation or atrial flutter ≥30 seconds.
2. Implanted pacemaker, cardiac defibrillator, cardiac loop recorder, or deep brain stimulator.
3. Likely to be poorly compliant or unreliable using home screening devices or with study follow-up requirements because of cognitive or other issues, or life expectancy <6 months due to concomitant disease.
4. Has a condition which in the opinion of the enrolling physician would not permit chronic treatment with oral anticoagulant therapy.
5. Patient already taking long-term oral anticoagulant therapy.
6. Known allergic reaction/intolerance to skin adhesives.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 856 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Detection of new atrial fibrillation or flutter | within 6 month from randomization
  Detection of new AF (atrial fibrillation or atrial flutter) within 6 months post-randomization, with AF defined as at least one episode of continuous AF lasting >5 minutes or AF documented on at least one 12-lead ECG or a convincing clinical diagnosis of AF based on reliable source documentation.

SECONDARY OUTCOMES:
Prescription of oral anticoagulation therapy | within 6 months from randomization
  Oral anticoagulant therapy use at 3 and 6 months post-randomization.
Primary endpoint detected by ECG patch monitor | within 6 months from randomization
  Among intervention group patients that meet the primary endpoint, detected by the ECG patch monitor, the following criteria will be analyzed:
  * time to first detection of AF >5 minutes
  * daily and total AF burden
  * average duration per AF episode.
Atrial fibrillation episodes of various durations (detection of any AF episode ≥30 seconds, ≥30 seconds to 5 minutes, >5 hours, and >24 hours (to facilitate comparison with other studies in the literature) | within 6 months from randomization
  Among intervention group patients, detection of any AF episode ≥30 seconds, ≥30 seconds to 5 minutes, >5 hours, and >24 hours (to facilitate comparison with other studies in the literature).
Adherence, tolerability and patient satisfaction with screening devices | within 6 months of randomization
  This is a composite outcome measured by the following:
  * Patient adherence with the screening devices (defined as the average number of monitoring days completed and reasons for non-adherence)
  * Patient satisfaction with the screening devices (as measured by user satisfaction surveys), - Tolerability of the ECG monitor (defined as the incidence of adverse skin reactions related to the adhesive patch).
Clinical outcome events | within 6 months from randomization
  A clinical outcome event will be defined as one of the following:
  * ischemic stroke
  * TIA
  * systemic embolism
  * major bleeding
  * intracranial hemorrhage
  * physician visits
  * hospitalizations
  * medication prescriptions. Clinical outcome events will be captured within 6 months post-randomization. The outcome is a composite measure.
Cost effectiveness of screening | within 6 months from randomization
  The cost effectiveness of screening is a composite outcome. The outcome will be measured by cost-effectiveness (cost per life year saved) and cost-utility (cost per quality adjusted life year (QALY) gained) of AF screening.
Detection of other (non-AF) clinically important arrhythmias | within 6 months from randomization
  Detection of other potentially clinically important non-AF arrhythmias: atrial tachycardia, pause >3 seconds, high-grade atrioventricular block (Mobitz type II or third-degree AV block), ventricular tachycardia, polymorphic ventricular tachycardia/ventricular fibrillation.
Sensitivity and specificity of Watch BP Home-A monitor ( false positive rate of a home AF-BP monitor (with ECG patch monitor as the gold standard). | within 6 months from randomization
  Estimated sensitivity, specificity and false positive rate of a home AF-BP monitor (with ECG patch monitor as the gold standard).

CONTACTS AND LOCATIONS:
Overall Officials: David J. Gladstone, MD PhD FRCPC, Principal Investigator — Sunnybrook Research Institute, University of Toronto
Locations (28):
- Canada (25):
  - Crowfoot Village Family Practice, Calgary, Alberta
  - Smith Clinic, Camrose, Alberta
  - Edmonton Oliver PCN, Edmonton, Alberta
  - Peaks to Praries PCN, Olds, Alberta
  - Henry Vlaar FP, Ayr, Ontario
  - LMC / Manna Research, Burlington, Ontario
  - Humber River FHT - Dixon Site, Etobicoke, Ontario
  - Halton Hills FHT, Georgetown, Ontario
  - Haileybury FHT, Haileybury, Ontario
  - Hamilton Medical Clinic, Hamilton, Ontario
  - Queen's Family Health Team, Kingston, Ontario
  - Ken Ng FP / Total Health Management, Markham, Ontario
  - St. Lawrence Medical Clinic, Morrisburg, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - OakMed FHT, Oakville, Ontario
  - Mark Robertson Family Practice, Owen Sound, Ontario
  - Garden City FHT, Saint Catherines, Ontario
  - Michael Kopp Family Practice / N Fung & M Kopp Medicine Professional Corporation, St. Catharines, Ontario
  - Health for All FHT, Stouffville, Ontario
  - Port Arthur Health Centre, Thunder Bay, Ontario
  - Keele Medical Place, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Mount Dennis Weston Health Centre, Toronto, Ontario
  - Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario
- Germany (3):
  - Goethe University Frankfurt am Main, Frankfurt am Main
  - Universitätsmedizin Göttingen, Göttingen
  - Hamburg University Medical School, Hamburg

REFERENCES:
- [Derived] Gladstone DJ, Wachter R, Schmalstieg-Bahr K, Quinn FR, Hummers E, Ivers N, Marsden T, Thornton A, Djuric A, Suerbaum J, von Grunhagen D, McIntyre WF, Benz AP, Wong JA, Merali F, Henein S, Nichol C, Connolly SJ, Healey JS; SCREEN-AF Investigators and Coordinators. Screening for Atrial Fibrillation in the Older Population: A Randomized Clinical Trial. JAMA Cardiol. 2021 May 1;6(5):558-567. doi: 10.1001/jamacardio.2021.0038. PMID 33625468
- See also: This website explains the SCREEN AF study and the C-SPIN network — http://www.cspin.ca/studies/piaaf/piaaf-home-screen-af/